CLINICAL TRIAL: NCT03985384
Title: Effect of Semaglutide on Coronary Atherosclerosis Plaque Progression in Type 2 Diabetics
Brief Title: Semaglutide Treatment On Coronary Progression
Acronym: STOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Matthew J. Budoff, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22174-01
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Active Comparator): Semaglutide 2mg/1.5 ml (1.34 mg/ml) Prefilled pen for SQ injection
  Interventions: Drug: Semaglutide 2 MG/1.5 ML Subcutaneous Solution
- Placebo (Placebo Comparator): Placebo 1.5 ml, pen-injector for SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide 2 MG/1.5 ML Subcutaneous Solution — Semaglutide 2 MG/1.5 ML Subcutaneous Solution
  Arms: Semaglutide
Drug: Placebo — Placebo 1.5 ml, pen-injector for SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to see the effect of the diabetes medicine Semaglutide on a condition called atherosclerosis. Atherosclerosis is a narrowing, blockage, or hardening of the arteries due to a build up of calcium. This study will look specifically at the arteries involving the heart.

DETAILED DESCRIPTION:
To determine the effects of semaglutide therapy on the morphology and composition of non-calcified coronary atherosclerotic plaque (NCP), including the progression of plaque volume.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with type 2 diabetes with a glycated hemoglobin level of 7.0% or more, drug naïve, or treated with oral agents and/or basal insulin. For patients on basal insulin at entry, the PI will consider dose reduction of basal insulin according to A1c and risk for hypoglycemia. Patients on SGLT-2 inhibitors may be screened but the agents must be discontinued at least 30 days prior to randomization.
* Age > 40 years of age at the time of the initial Screening visit (V1) with a diagnosis of T2DM in accordance with American Diabetes Association (ADA) guidelines and with at least one cardiovascular risk factor (hypertension, high cholesterol, family history of premature heart disease or past/current smoking) or prior ASCVD (prior stroke, TIA, claudication, coronary artery disease)
* Willingness to participate in the study and ability to sign informed consent
* In the investigator's opinion subjects are willing and likely able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures whether or not they receive investigational product for the duration of the trial.

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis.
* Current use of GLP-1-receptor agonists or use of a GLP-1 receptor agonist within 3 mos. of screening.
* Current Use of SGLT-2 inhibitors within 30 days of screening
* Subjects on prandial insulin or using an insulin pump or pramlintide.
* Any clinically significant malabsorption condition.
* History of one or more severe hypoglycemic episodes within 6 months of Screening (V1) or a severe hypoglycemic episode occurring during the interval between the Screening visit (V1) and randomization.
* Subjects experiencing a cardiovascular event (e.g., myocardial infarction or stroke) or undergoing coronary angioplasty or peripheral intervention procedure between the Screening visit (V1) and randomization.
* Recent ASCVD Event (stroke, heart attack, ACS or revascularization) within 3 months (90 days) of the screening visit (VI).
* Subjects undergoing any cardiovascular surgery (e.g., valvular surgery) within 3 months (90 days) of the Screening visit (V1).
* Subjects with any planned coronary revascularization or peripheral intervention procedure or other cardiovascular surgery.
* Subjects with New York Heart Association (NYHA) Class III or IV heart failure at the Screening visit (V1).
* Renal insufficiency (calculated creatinine clearance of <50 ml per minute, MDRD equation).
* AST or ALT >2 X the upper limit of normal (ULN) at the Screening visit (V1), or a total bilirubin >1.5 X the ULN unless the subject has a history of Gilbert's.
* Weight in excess of 325 pounds
* Resting hypotension (systolic blood pressure of <90mmHg) or resting hypertension (systolic blood pressure of >170mmHg or diastolic blood pressure of >110 mmHg) or the treating physician is allowed to adjust background blood pressure medication(s) to lower blood pressure values in order for the subject to be re-assessed for enrollment eligibility.
* Subject has a history of malignancy ≤5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.

Note (1) A subject with a history of malignancy >5 years prior to signing informed consent should have no evidence of residual or recurrent disease.

Note (2) a subject with any history of melanoma, leukemia, lymphoma, or renal cell carcinoma is excluded.

* At randomization, subject has developed a new medical condition, suffered a change in status of an established medical condition, developed a laboratory or ECG abnormality, or required a new treatment or medication during the pre-randomization period which meets any previously described trial exclusion criterion or which, in the opinion of the investigator, exposes the subject to risk by enrolling in the trial.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality at the Screening visit (V1) that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
* Subjects with known allergy to iodinated contrast material
* Subject is pregnant or breast-feeding, or is expecting to conceive during the trial, including 35 days following the last dose of blinded investigational product.
* Females of childbearing potential must use adequate contraceptive methods.
* Participation in other studies involving investigational drug (s) (Phases 1-4) within 30 days before the Screening visit (V1) and/or during trial participation.
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC)
* Personal history of non-familial medullary thyroid carcinoma.
* Known or suspected hypersensitivity to trial products.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Rate of change in non-calcified plaque volume | 12 months
  Rate of change in non-calcified plaque volume

SECONDARY OUTCOMES:
Rate of change in total plaque volume | 12 months
  Rate of change in total plaque volume

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Budoff, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California, United States